CLINICAL TRIAL: NCT06983444
Title: Bipolar Trans Urethral Resection of the Prostate (TURP) Versus Bipolar Enucleation of the Prostate in Treatment of Benign Prostatic Hyperplasia (BPH): A Prospective Randomized Comparative Clinical Study
Brief Title: Bipolar Resection vs Enucleation of Prostate
Acronym: TURP vs BiTUEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelfattah Hamed Abdelraheem, Assistant Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endoscopic surgery prostate
Record Dates: First submitted 2025-04-29; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Benign Prostatic Hyperplasia (BPH) Requiring Surgical Resection; Benign Prostatic Hyperplasia With Outflow Obstruction; Benign Prostatic Hyperplasia With Symptomatic Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia With Lower Urinary Tract Symptoms
Keywords: TURP; TUEP; BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: A comparison between TURP and Bipolar enucleation of prostate allows us to investigate the true benefits and safety of each modality.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transurethral resection of prostate (Active Comparator): Transurethral resection of prostate (TURP) will be performed under spinal or general anesthesia as per usual care.
  Interventions: Procedure: TURP
- Transuretheral enucleation of prostate (Active Comparator): Transurethral enucleation of prostate (TUEP) will be performed under spinal or general anesthesia as per usual care.
  Interventions: Procedure: TUEP

INTERVENTIONS:
Procedure: TURP — Using bipolar loop diathermy via cystoscopy, excess prostate tissue is resected piecemeal to remove obstruction to the prostatic urethra due to BPH.
  Other Names: Transurethral resection of prostate; Bipolar TURP
  Arms: Transurethral resection of prostate
Procedure: TUEP — Using bipolar enucleation loop diathermy via cystoscopy, to anatomically enucleate prostate.
  Other Names: Transurethral enucleation of prostate; Bipolar TUEP; Anatomical endoscopic enucleation of prostate; AEEP
  Arms: Transuretheral enucleation of prostate

SUMMARY:
The aim of this study is to evaluate efficacy and safety of transurethral resection of the prostate and bipolar enucleation of the prostate.

DETAILED DESCRIPTION:
Endoscopic management of benign prostatic hyperplasia (BPH), monopolar transurethral resection of the prostate (TURP) has been the gold standard for many years.

Despite its promising efficacy in treating BPH, TURP is associated with a risk of significant complications and clinical limitations, including life-threatening events such as transurethral resection (TUR) syndrome, as well as high cost due to long hospital stay, long catheterization time and difficulty in management of large sized prostate so alternative surgical approaches have been explored.

Minimally invasive approaches achieve equal efficiency to standard resection, but with a more favorable safety and less complications.

Anatomical enucleation of the prostate using Bipolar or Laser-based approaches such as holmium laser have been introduced with success and the efficacy and safety of these procedure has led to the integration into several international guidelines.

Early results of bipolar enucleation resemble those reported for holmium laser procedure, Bipolar transurethral enucleation of the prostate was at least equally effective, and showed less complications, good hemostatic control and both shorter catheterization time and hospital stay than old standard procedure.

A comparison between TURP and Bipolar enucleation of prostate allows us to investigate the true benefits and safety of each modality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lower urinary tract symptoms (LUTS) due to BPH.
2. Patients with international prostate score system (IPSS) more than 8.
3. Patients with maximal urinary flow rate (Qmax) less than 10ml/second.
4. Patients with Prostatic volume (60 - 100 gm).
5. Patient with indication for surgical intervention.
6. Patient age (50-80 years old)

Exclusion Criteria:

1. Prostatic cancer.
2. Bladder cancer.
3. Urethral stricture.
4. Neurogenic bladder.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patient with BPH
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Catheter and lower urinary tract symptoms free after Bipolar Transurethral resection of prostate (TURP) versus Bipolar Transurethral enucleation of prostate (TUEP) in patient with BPH with lower urinary tract symptoms | at least 6 months up to one year
  To determine number of patients in each group that will be Catheter and lower urinary tract symptoms free with changes in IPPS < 20 score after intervention and follow up at 1 month, 3 months and 6 months.

SECONDARY OUTCOMES:
Operative time in minutes in each group of intervention | 60 - 90 minutes for each group of intervention
  To determine operative time in minutes in each group of intervention
Compare complication rate of TURP versus TUEP | at least 6 months up to one year
  To determine the percentage and severity of complications after each intervention (according to the Clavien-Dindo classification).
  * Minimum score is class I: No intervention needed
  * Maximum score is class V: Death of a patient
Cost effectiveness of TURP versus TUEP in achieving catheter-free rates in BPH patients with urinary retention | at least 6 months up to one year
  To determine the cost required to achieve catheter free patients for each intervention (including hospitalization, anesthetic costs, equipment, consumables, etc)
Compare patient reported symptom measures by IPSS questionnaire after TURP versus TUEP | at least 6 months up to one year
  sing International prostate symptom score (IPSS) questionnaire to determine patient reported symptom measure after each intervention
  minimal score: 0, maximum score is 35 higher score means worse outcome
Compare patient reported symptom measures by Michigan Incontinence Symptom Index (M-ISI) questionnaire after TURP versus TUEP | at least 6 months up to one year
  Using the Michigan Incontinence Symptom Index (M-ISI) questionnaire to determine patient reported symptom measure after each intervention
  * Minimum score: 1
  * Maximum score: 12
  * The higher the score means worse outcome
Compare patient reported symptom measures by IIEF-5 questionnaire after TURP versus TUEP | at least 6 months up to one year
  Using the International index of erectile function- 5 items (IIEF-5) questionnaire to determine patient reported symptom measure after each intervention
  minimum score: 1, maximum score: 25 higher score means better outcome
Compare patient reported quality of life by SF-12 questionnaire after TURP versus TUEP | at least 6 months up to one year
  sing the Short Form 12 (SF-12) questionnaire to determine patient reported quality of life measures after each intervention
  minimum score: 0, maximum score: 100 higher score means better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Yuan P, Ma D, Gao X, Wei C, Liu Z, Li R, Wang S, Liu J, Liu X. Efficacy and safety of enucleation vs. resection of prostate for treatment of benign prostatic hyperplasia: a meta-analysis of randomized controlled trials. Prostate Cancer Prostatic Dis. 2019 Dec;22(4):493-508. doi: 10.1038/s41391-019-0135-4. Epub 2019 Feb 28. PMID 30816336
- [Background] Seitz M, Sroka R, Gratzke C, Schlenker B, Steinbrecher V, Khoder W, Tilki D, Bachmann A, Stief C, Reich O. The diode laser: a novel side-firing approach for laser vaporisation of the human prostate--immediate efficacy and 1-year follow-up. Eur Urol. 2007 Dec;52(6):1717-22. doi: 10.1016/j.eururo.2007.06.028. Epub 2007 Jun 26. PMID 17628326
- [Background] Bachmann A, Schurch L, Ruszat R, Wyler SF, Seifert HH, Muller A, Lehmann K, Sulser T. Photoselective vaporization (PVP) versus transurethral resection of the prostate (TURP): a prospective bi-centre study of perioperative morbidity and early functional outcome. Eur Urol. 2005 Dec;48(6):965-71; discussion 972. doi: 10.1016/j.eururo.2005.07.001. Epub 2005 Jul 18. PMID 16126327
- [Background] Gilling PJ, Wilson LC, King CJ, Westenberg AM, Frampton CM, Fraundorfer MR. Long-term results of a randomized trial comparing holmium laser enucleation of the prostate and transurethral resection of the prostate: results at 7 years. BJU Int. 2012 Feb;109(3):408-11. doi: 10.1111/j.1464-410X.2011.10359.x. Epub 2011 Aug 23. PMID 21883820
- [Background] Arcaniolo D, Manfredi C, Veccia A, Herrmann TRW, Lima E, Mirone V, Fusco F, Fiori C, Antonelli A, Rassweiler J, Liatsikos E, Porpiglia F, De Sio M, Autorino R; EAU Section of Uro-Technology (ESUT) Research Group. Bipolar endoscopic enucleation versus bipolar transurethral resection of the prostate: an ESUT systematic review and cumulative analysis. World J Urol. 2020 May;38(5):1177-1186. doi: 10.1007/s00345-019-02890-9. Epub 2019 Jul 25. PMID 31346761
- [Background] Ho HS, Yip SK, Lim KB, Fook S, Foo KT, Cheng CW. A prospective randomized study comparing monopolar and bipolar transurethral resection of prostate using transurethral resection in saline (TURIS) system. Eur Urol. 2007 Aug;52(2):517-22. doi: 10.1016/j.eururo.2007.03.038. Epub 2007 Mar 28. PMID 17416453